CLINICAL TRIAL: NCT06981078
Title: A Phase 2b Randomized, Double-blind, Placebo-controlled, Parallel-Group Study to Assess Efficacy and Safety of Verekitug (UPB-101) in Participants With Moderate-to-Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study to Assess the Efficacy and Safety of Verekitug in Participants With COPD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Upstream Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UPB-CP-06; 2025-520488-42-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-09; First posted 2025-05-20 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Verekitug; UPB-101; Chronic Obstructive Pulmonary Disease; Emphysema; Chronic Bronchitis; Thymic Stromal Lymphopoetin Receptor; Lung Inflammation; Biologic; Monoclonal Antibody; VENTURE
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Verekitug (UPB-101) 100 mg and Placebo (Experimental): Participants will receive 0.5 milliliter (mL) of the formulated solution (containing 100 milligrams [mg] of verekitug [UPB-101]) and 2.0 mL of matching placebo subcutaneously in two separate injections every 12 weeks up to Week 96.
  Interventions: Drug: Verekitug; Other: Placebo
- Verekitug (UPB-101) 400 mg and Placebo (Experimental): Participants will receive 2.0 mL of the formulated solution (containing 400 mg of verekitug [UPB-101]) and 0.5 mL of matching placebo subcutaneously in two separate injections every 24 weeks up to Week 96. Participants will also receive 2.0 mL and 0.5 mL of matching placebo subcutaneously in two separate injections at Weeks 12, 36, 60 and 84 visits.
  Interventions: Drug: Verekitug; Other: Placebo
- Placebo (Placebo Comparator): Participants will receive 0.5 mL of matching placebo and 2.0 mL of matching placebo subcutaneously in two separate injections every 12 weeks up to Week 96.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Verekitug — Verekitug (UPB-101) formulated solution
  Other Names: UPB-101
  Arms: Verekitug (UPB-101) 100 mg and Placebo; Verekitug (UPB-101) 400 mg and Placebo
Other: Placebo — Matching Placebo to Verekitug (UPB-101)

SUMMARY:
The purpose of this study is to assess the efficacy and safety of verekitug (UPB-101) in participants with moderate-to-severe Chronic Obstructive Pulmonary Disease (COPD), an inflammatory lung disease.

DETAILED DESCRIPTION:
This is a global, multicenter study to assess the efficacy, safety, and tolerability of verekitug in participants with moderate-to-severe COPD. Adult participants are planned to be enrolled and will be allocated randomly in a 1:1:1 ratio to one of two dose levels of verekitug or placebo, in addition to their COPD background medications. The study consists of a screening period of approximately 4 weeks; treatment periods of between 60 weeks and up to 108 weeks; and a follow-up period, with the end-of-study visit 16 weeks after last dose.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of COPD for >12 months.
* Current or former smokers with a smoking history of 10 pack-years or more.
* Post-bronchodilator FEV1/ Forced Vital Capacity (FVC) ratio <0.70 and predicted post-bronchodilator FEV1 >30% and ≤80%.
* Modified Medical Research Council dyspnea scale Grade ≥2.
* Background triple therapy (Inhaled Corticosteroid [ICS], Long-Acting Beta Agonist [LABA], Long-Acting Muscarinic Antagonist [LAMA]) for 3 months before randomization with a stable dose of medications for 1 or more months prior to Visit 1.
* Are ≥80% compliant with background therapy during the screening period.

Exclusion Criteria:

* Moderate or severe exacerbation of COPD within 4 weeks prior to or during the screening period.
* Respiratory tract infection within 4 weeks prior to or during the screening period.
* Treatment with oxygen of >4 liters/minute. Nocturnal oxygen use for sleep apnea is allowed.
* Systemic or biologic immunosuppressant therapy to treat inflammatory disease or autoimmune disease within 24 weeks or 5 half-lives prior to Visit 1, whichever is longer, with the exception of oral corticosteroids. Treatment with cyclophosphamide and rituximab within 12 months of Visit 1.
* Current diagnosis of asthma according to the 2023 Global Initiative for Asthma guidelines or other accepted guidelines
* History or evidence of a clinically meaningful pulmonary condition other than COPD (e.g., pulmonary fibrosis, sarcoidosis, interstitial lung disease, pulmonary hypertension, bronchiectasis, Churg-Strauss Syndrome) or another diagnosed pulmonary or systemic disease associated with elevated peripheral eosinophil counts.
* Chronic hypercapnia requiring Bilevel Positive Airway Pressure (BiPAP). Participants requiring BiPAP periodically for an acute COPD exacerbation are not excluded.
* Any of the following in the previous 6 months prior to Visit 1: acute myocardial infarction, transient ischemic attack or stroke, hospitalization for any cardiovascular or cerebrovascular event, pulmonary embolism, deep vein thrombosis and cardiac arrhythmias including paroxysmal (e.g., intermittent). Participants with persistent atrial fibrillation as defined by continuous atrial fibrillation for at least 6 months and controlled with a rate control strategy (i.e., selective beta blocker, calcium channel blocker, pacemaker placement, digoxin or ablation therapy) and stable appropriate level of anticoagulation for at least 6 months may be considered for inclusion.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of moderate or severe COPD exacerbation events | From Day 1 (Baseline) up to Week 108

SECONDARY OUTCOMES:
Change in pre-bronchodilator forced expiratory capacity in 1 second (FEV1) | From Day 1 (Baseline) to Week 60
Annualized rate of severe COPD exacerbation events | From Day 1 (Baseline) up to Week 108
Change in St. George's Respiratory Questionnaire (SGRQ) total score | From Day 1 (Baseline) to Week 60
Proportion of participants with SGRQ improvement of >4 points | At Week 60
Incidence of treatment-emergent adverse events and serious adverse events | From Day 1 (Baseline) up to Week 112

CONTACTS AND LOCATIONS:
Overall Officials: Justin Salciccioli, MD, Study Director — Upstream Bio
Locations (322):
- United States (32):
  - Quality of Life Med Research, Tucson, Arizona
  - Kern Research Inc., Bakersfield, California
  - PulmoCrit Associates, Encino, California
  - Torrance Clinical Research Institute, Lomita, California
  - Dream Team Clinical Research, Pomona, California
  - Apex Clinical Research, San Diego, California
  - Allianz Research Institute, Westminster, California
  - Allianz Research Institute, Aurora, Colorado
  - D&H Doral Research Center, LLC, Doral, Florida
  - Qway Research, LLC, Hialeah, Florida
  - Finlay Medical Research, Miami, Florida
  - Research Institute of South Florida, Miami, Florida
  - Florida Institute for Clinical Research,LLC, Orlando, Florida
  - Velocity Clinical Research-Savannah - Internal Medicine, Savannah, Georgia
  - Christie Clinic, LLC, Champaign, Illinois
  - The Iowa Clinic, West Des Moines, Iowa
  - Velocity Clinical Research-Rockville, Rockville, Maryland
  - Chesapeake Clinical Research, Inc, White Marsh, Maryland
  - HealthPartners, Saint Paul, Minnesota
  - American Health Research, Inc., Charlotte, North Carolina
  - Velocity Clinical Research, Anderson, Anderson, South Carolina
  - SleepMed Inc., Columbia, South Carolina
  - Velocity Clinical Research, Gaffney, Greenville, South Carolina
  - Velocity Clinical Research, Spartanburg - Pulmonology, Spartanburg, South Carolina
  - Velocity Clinical Research- Union, Union, South Carolina
  - Elligo Health Research, Inc., Austin, Texas
  - El Paso Pulmonary Association, El Paso, Texas
  - Victorium Clinical Research, Houston, Texas
  - Synergy Groups Medical LLC, Houston, Texas
  - Metroplex Pulmonary and Sleep Center, McKinney, Texas
  - Synergy Groups Medical LLC, Missouri City, Texas
  - Velocity Clinical Research - Suffolk, Suffolk, Virginia
- Argentina (24):
  - IADIN - Research, Buenos Aires, Buenos Aires
  - Fundacion CIDEA, Buenos Aires, Buenos Aires
  - Hosp Zonal Espec en Agudos y Cronicos "Dr. A. A. Cetrangolo" - Intensive Respiratory Care, Buenos Aires, Buenos Aires
  - CARE - Centro de Alergia y Enfermedades Respiratorias, Buenos Aires, Buenos Aires
  - Consultorios Médicos Dr. Doreski, Buenos Aires, Buenos Aires
  - Centro Medico CIMEL CHAHIN CHAHIN, Lanús, Buenos Aires
  - Centro de Investigaciones Medicas Mar del Plata - internal medicine, Mar del Plata, Buenos Aires
  - Fundacion Enfisema, Mar del Plata, Buenos Aires
  - Clinica Privada Monte Grande S.A, Monte Grande, Buenos Aires
  - IERIM-Instituto de Enfermedades Respiratoria e Investigacion Médica, San Juan Bautista, Buenos Aires
  - CEMER, Vicente López, Buenos Aires
  - Cli-nica Adventista Belgrano - investigacion, Buenos Aires, Buenos Aires F.D.
  - Clinica Colombo - Cardiology, Córdoba, Córdoba Province
  - Centro de Medicina Respiratoria, Concepción del Uruguay, Entre Ríos Province
  - Framingham Centro Medico, La Plata, Entre Ríos Province
  - Hospital Español de Mendoza, Godoy Cruz, Mendoza Province
  - Fundacion Scherbovsky, Mendoza, Mendoza Province
  - Centro Respiratorio Quilmes, Buenos Aires, Quilmes
  - National University of Cordoba - Rusculleda Foundation - Instituto DAMIC, Córdoba, Río Negro Province
  - Fundacion Estudios Clinicos (FECLIN), Rosario, Santa Fe Province
  - Instituto Médico Fundación Grupo Colaborativo Rosario Invest, Rosario, Santa Fe Province
  - Ibamedica, Santa Fe, Santa Fe Province
  - Investigaciones en Patologias Respiratorias, San Miguel de Tucumán, Tucumán Province
  - Centro Medico Privado de Reumatologia - Servicio de Reumatología, San Miguel de Tucumán, Tucumán Province
- Bulgaria (22):
  - Medical Center Pulmo-2018 EOOD, Haskovo, Haskovo
  - Medical Center Medconsult Pleven, Lovech branch, Lovech, Lovech
  - MEDICAL CENTER HERA EOOD; Office of Pulmonology and Phtisiatrics, Montana, Montana
  - SHLTTRPD "Sveta Petka Balgarska" EOOD, Velingrad, Pazardzhik
  - Specialized Hospital For Active Treatment Of Pulmonary Diseases Sv.Panteleymon EOOD, Dupnitsa, Pernik
  - Dr. Filip Shterev IAPSMCPP EOOD, Plovdiv, Plovdiv
  - Medical Center Etika Ambulatory For Specialized Outpatient Medical Care OOD, Plovdiv, Plovdiv
  - Multiprofile Hospital for Active Treatment "St. Panteleimon "- Plovdiv, Plovdiv, Plovdiv
  - Medical Center Prolet EOOD - Pulmonary, Allergy Diseases, Rousse, Ruse
  - Specialized Hospital For Active Treatment Of Pneumo-Phthisiatric Diseases Dr. Dimitar Gramatikov-Ruse EOOD, Rousse, Ruse
  - Diagnostic consultative center 1 -Sliven, Sliven, Sliven
  - MHAT Sliven to MMA Sofia, Sliven, Sliven
  - Medical Center Excelsior OOD, Base 2, Sofia, Sofia
  - Acibadem City Clinic Tokuda University Hospital EAD, Sofia, Sofia
  - First Multiprofile Hospital for Active Treatment - Sofia, Sofia, Sofia-Grad
  - Specialized Hospital For Active Treatment Of Pulmonary Diseases - Sofia EOOD, Sofia, Sofia-Grad
  - National Multiprofile Transport Hospital (NMTB) - Internal Diseases, Sofia, Sofia-Grad
  - Medical Center Excelsior OOD, Base 1, Sofia, Sofia-Grad
  - Medical Center Hera, Sofia, Sofia-Grad
  - DCC Convex EOOD, Sofia, Sofia-Grad
  - Medical Center for Outpatient Care Preventsia 2000, Stara Zagora, Stara Zagora
  - Medical Center - Zdrave1, Kozloduy, Vratsa
- Chile (6):
  - Bioreuma, Concepción, Maule Region
  - Centro Investigación Maule, Talca, Maule Region
  - Ctro Respiratorio Integral CENRESIN, Quillota, Región de Valparaíso
  - Centro de Investigación de Enfermedades Respiratorias e Inmunológicas, Viña del Mar, Región de Valparaíso
  - Centro de Investigaciones Clínicas Viña del Mar, Viña del Mar, Región de Valparaíso
  - Clinica Fundacion Medica San Cristobal, Vitacura, Santiago Metropolitan
- Czechia (11):
  - EDUMED, s.r.o, Broumov, Královéhradecký kraj
  - Plicni ambulance Alveolus s.r.o., Poruba, Moravskoslezský kraj
  - MEDICON a.s. - Plicni oddeleni, Prague, Praha, Hlavní Mesto
  - Privatni plicni ambulance, s.r.o., Prague, Praha, Hlavní Mesto
  - Plicni ambulance Rokycany, Rokycany, Rokycany
  - MUDr. Pavlisova Ilona s.r.o., Miroslav, South Moravian
  - Ordinace pro TBC a respiracni nemoci - Ordinace pro TBC a resp.nem., Strakonice, Strakonice
  - MUDr. I. Cierna Peterova s.r.o., Brandýs nad Labem, Stredoceský Kraj
  - Plicni ambulance Kralupy s.r.o., Kralupy nad Vltavou, Stredoceský Kraj
  - Plicni stredisko Teplice s.r.o. - Plicni ordinace, Teplice, Ústecký kraj
  - Pneumologie Varnsdorf s.r.o., Varnsdorf, Ústecký kraj
- Georgia (8):
  - LTD "High Technology Hospital Medcenter", Batumi, Adjara
  - LTD Clinic Rustavi, Rustavi, Hvemo Kartli
  - A. Aladashvili clinic LLC, Tbilisi, K'alak'i T'bilisi
  - LTD "Israel-Georgian Medical Research Clinic Healthycore", Tbilisi, K'alak'i T'bilisi
  - Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic, Tbilisi, K'alak'i T'bilisi
  - Center of Allergy and Immunology - Allergy/Immunology-Reumatology, Tbilisi, K'alak'i T'bilisi
  - Ltd Diacor, Tbilisi, K'alak'i T'bilisi
  - LTD MARNECOR - Internal Medicine, Marneuli, Kvemo Kartli
- Germany (20):
  - Gemeinschaftspraxis Rolke / Rückert, Aschaffenburg, Bavaria
  - Pneumologie, Schlafmedizin und Onkologie am Diako, Augsburg, Bavaria
  - CIMS Studienzentrum Bamberg, Bamberg, Bavaria
  - Asklepios Lungenklinik Gauting GmbH - Zentrum für Pneumologie und Thoraxchirurgie, München, Bavaria
  - MECS GmbH, Cottbus, Brandenburg
  - ME Clinical Respiratory Research, Hamburg, Hamburg
  - Pneumostudien Darmstadt GmbH, Darmstadt, Hesse
  - IKF Pneumologie GmbH & Co. KG, Frankfurt am Main, Hesse
  - Ballenberger, Freytag, Wenisch, Neu-Isenburg, Hesse
  - Pneumologische Praxis und Schlaflabor - Lutz Volgmann, Hanover, Lower Saxony
  - Studienzentrum Dr.med. Christian Schlenska - Pneumologie/Allergologie/Innere Medizin, Peine, Lower Saxony
  - Framol-Med GmbH, Rheine, North Rhine-Westphalia
  - Gemeinschaftspraxis Franz, Weber, Witten, North Rhine-Westphalia
  - IKF Pneumologie GmbH & Co. KG, Mainz, Rhineland-Palatinate
  - Pneumologicum-Halle - Pulmonary, Halle, Saxony-Anhalt
  - Velocity Clinical Research Germany GmbH, Lübeck, Schleswig-Holstein
  - Studienpraxis Berlin-Brandenburg, Berlin, State of Berlin
  - Lungenpraxis Hohenzollerndamm, Berlin, State of Berlin
  - Velocity Clinical Research Germany GmBH, Berlin, State of Berlin
  - MECS Research GmbH, Berlin, State of Berlin
- Hungary (12):
  - Infer-Med Kft., Pécs, Baranya
  - Bekes Varmegyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula, Bekes County
  - Koch Róbert Kórház és Rendel?intézet, Edelény, Borsod-Abauj Zemplen county
  - ClinExpert Kft., Budapest, Budapest
  - Pulmo Protect Kft., Budapest, Budapest
  - Kek Pont Aquagyogyaszat Kft., Kecskemét, Bács-Kiskun county
  - Aranyklinika Kft, Bordány, Csongrád megye
  - Debreceni Egyetem Klinikai Központ - Tüdőgyógyászati Klinika, Debrecen, Debrecen
  - Szalay Janos Rendelointezet, Hajdúnánás, Hajdú-Bihar
  - Puspokladanyi Egeszsegugyi Szolgaltato Nonprotfit Kft, Püspökladány, Heves County
  - Erzsebet Gondozohaz Kft., Gödöllő, Pest County
  - Farkasgyepui Tudogyogyintezet, Farkasgyepű, Veszprém megye
- India (14):
  - Astar Prime Hospitals - Internal Medicine, Hyderabad, Andhra Pradesh
  - A.C. Subba Reddy Government Medical College (ACSR) - Pulmonary, Nellore, Andhra Pradesh
  - Siddhartha Medical College, Vijayawada, Andhra Pradesh
  - Medanta Medicity, Gurgaon, Haryana
  - Pandit Bhagwat Dayal Sharma Post Graduate Institute of Medical Sciences (PGIMS) - Pandit Bhagwat Dayal Sharma, Rohtak, Haryana
  - Rajarshi Chhatrapati Shahu Maharaj (RCSM) Government Medical College & CPR Hospital, Kolhāpur, Maharashtra
  - Shree Hospital & Critical Care Centre, Nagpur, Maharashtra
  - Sir Ganga Ram Hospital (SGRH) - Gastroenterology and Hepatology, New Delhi, National Capital Territory of Delhi
  - Fortis Hospital Mohali, Mohali, Punjab
  - S.P Medical College and Group of Hospitals, Bikaner, Bikaner, Rajasthan
  - King George's Medical University, Lucknow, Uttar Pradesh
  - Shri Mahant Indiresh Hospital, Dehradun, Uttarakhand
  - JNMC, Belgaum, West Bengal
  - NRS Medical College, Kolkata, West Bengal
- Ireland (7):
  - Cork University Hospital, Cork, Cork
  - St Vincent's University Hospital, Dublin, Dublin
  - Connolly Hospital, Dublin, Dublin
  - Tallaght University Hospital, Tallaght, Dublin
  - University College Hospital Galway - Pulmonology, Galway, Galway
  - University Hospital Limerick, Limerick, Limerick
  - Our Lady of Lourdes Hospital, Drogheda, Louth
- Latvia (5):
  - Daugavpils Regional Hospital, Daugavpils, Daugavpils
  - Veselibas Centru apvieniba AS, Dubultu poliklinika, Jūrmala, Jūrmala
  - Liepaja Regional Hospital, Liepāja, Liepāja
  - Pauls Stradins Clinical University Hospital - Center of Lung Diseases, Riga, Rīga
  - SIA "Profesora Skrides Sirds klīnika", Riga, Rīga
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas, Kaunas County
  - Lithuanian University of Health Sciences Kaunas Hospital, Kaunas, Kaunas County
  - Republic Klaipeda Hospital, Klaipėda, Klaipėda County
- Malaysia (5):
  - Institut Perubatan Respiratori, Kuala Lumpur, Kuala Lumpur
  - Universiti Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Thomson Hospital Kota Damansara, Petaling Jaya, Selangor
  - Universiti Teknologi MARA, Shah Alam, Selangor
- Mexico (5):
  - Instituto Jalisciense de Metabolismo, SC - Research, Guadalajara, Jalisco
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez - CIPTIR, Monterrey, Nuevo León
  - Unidad Inv Clinica Medicina, Monterrey, Nuevo León
  - Centro Respiratorio de México, México, State of Mexico
  - Phylasis Clinicas Research S de RL de CV; Sucursal Toluca, Toluca, State of Mexico
- Philippines (9):
  - Marilao Saint Michael Family Hospital, Inc. - Research Room, Marilao, Bulacan
  - CARE Clinical Trial Group Inc., Dasmariñas, Cavite
  - De Asis Medical Clinic (Norzel Medical and Diagnostic Clinic), Cebu, Cebu
  - Perpetual succour hospital of Cebu INC, Cebu, Cebu
  - Iloilo Doctors' Hospital Inc., Iloilo City, Iloilo
  - St. Paul's Hospital of Iloilo Inc. - Pulmonology, Iloilo City, Iloilo
  - Health Cube Medical Clinics, Mandaluyong, National Capital Region
  - Asian Hospital and Medical Center - Medicine, Muntinlupa, National Capital Region
  - Lung Center Of the Philippines - Medicine, Quezon City, National Capital Region
- Poland (15):
  - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz, Greater Poland Voivodeship
  - Specjalistyczna Przychodnia Lekarska Alergo - Med Sp. z o.o., Poznan, Greater Poland Voivodeship
  - Centrum Medyczne ALL-MED, Krakow, Lesser Poland Voivodeship
  - Pratia MCM Kraków, Krakow, Lesser Poland Voivodeship
  - Clinical Best Solutions, Lublin, Lubusz Voivodeship
  - Twoja Przychodnia Nowosolskie Centrum Medyczne Sp. z o. o., Nowa Sól, Lubusz Voivodeship
  - Velocity Skierniewice Sp. z o.o., Skierniewice, Lódzkie
  - RCMed Oddzial Sochaczew, Sochaczew, Masovian Voivodeship
  - Prywatny Gabinet Lekarski, Rzeszów, Podkarpackie Voivodeship
  - EMED Centrum Uslug Medycznych Ewa Smialek, Rzeszów, Podkarpackie Voivodeship
  - Centrum Medycyny Oddechowej, Mroz Spolka Jawna, Bialystok, Podlaskie Voivodeship
  - ClinicMed Daniluk, Nowak Sp. Komandytowa, Bialystok, Podlaskie Voivodeship
  - Uniwersyteckie Centrum Kliniczne - Klinika Alergologii, Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne Pratia Katowice, Katowice, Warmian-Masurian Voivodeship
  - Twoja Przychodnia Szczecinskie Centrum Medyczne Sp. z o. o., Szczecin, West Pomeranian Voivodeship
- Romania (12):
  - Centrul Medical de Diagnostic si Tratament Ambulator Neomed - Multiple Specialties, Brasov, Brașov County
  - Centrul Medical Sana, Bucharest, București
  - Medsana CM Cotroceni Pulmonology, Bucharest, București
  - Rimmed Centru Medical Pulmonology, Bucharest, București
  - Anima Specialty Medical Services, Bucharest, București
  - CM Pneumologie Dr Mincu Bogdan, Cluj-Napoca, Cluj
  - Sp Pneumoftizio Leon Daniello CJ, Cluj-Napoca, Cluj
  - Sp.Clinic Pneumo Constanta Pulmon 2, Palazu Mare, Constanța County
  - Angisan Grup, Bragadiru, Ilfov
  - Fundatia Dr. Victor Babes, Bucuresti, Ilfov
  - Clintrial Medical Center, Dobrosloveni, Olt
  - Sp Dr Victor Babes Timisoara Pulmon, Timișoara, Timiș County
- Serbia (12):
  - Military Medical Academy, Belgrade, Belgrade
  - MSB General hospital - Clinical Research Center, Belgrade, Belgrade
  - Municipal Institute for Lung Diseases and Tuberculosis - Allegology and Clinical Immunology, Belgrade, Belgrade
  - Clinical Hospital Center "Bezanijska Kosa" Clinic for Intern - Pulmology, Belgrade, Belgrade
  - University Clinical Center of Serbia, Clinic for Pulmonology- IV Department of General Pulmonology, Belgrade, Belgrade
  - General Hospital Valjevo - Department for Pulmology, Valjevo, Kolubarski okrug
  - Clinical Center Nis,Clinic for Pulmonary Diseases - Pulmonary Diseases & Tuberculosis, Niš, Nišavski okrug
  - General Hospital Jagodina/Internal Medicine department, Jagodina, Pomoravski okrug
  - nstitute for Pulmonary Diseases of Vojvodina, Clinic for Pulmonary Oncology, Kamenitz, Vojvodina
  - General Hospital Uzice, Department for Pulmonology, Užice, Zlatiborski okrug
  - Polyclinic Aleksandar Rahec Radojevic, Čačak, Šumadijski Okrug
  - University Clinical Center of Kragujevac, Clinic for Pulmonology, Kragujevac, Šumadijski Okrug
- Slovakia (8):
  - FNsP F.D.R. Banska Bystrica - Pneumologie a ftizeologie, Banská Bystrica, Banská Bystrica Region
  - PAFA, s.r.o., Bratislava, Bratislava Region
  - Pneumomed s.r.o. - Pneumo-Alergo Centrum, Bratislava, Bratislava Region
  - MEDEKA s.r.o. - Pneumologia a ftizeologia, Košice, Košice Region
  - Plucna ambulancia Hrebenar s.r.o., Spišská Nová Ves, Košice Region
  - ZAPA JJ s.r.o. - Pneumologia a ftizeologia, Levice, Nitra Region
  - DIONEA, s.r.o. - Ambul. pneumologie, Nové Zámky, Nitra Region
  - INSPIRO s.r.o. - MUDr. Golubov Alexander - Pneumologia a ftizeologia, Humenné, Presov
- South Africa (10):
  - MeDiNova Merc Clinical Research, Welkom, Free State
  - WWCT -Lakeview Hospital, Benoni, Gauteng
  - Ryexo Clinical Research -Wilgers, Pretoria, Gauteng
  - FCRN Clinical Trial Centre, Vereeniging, Gauteng
  - Practice Dr Visvakuren Naidoo - Clinical Trials, Durban, KwaZulu-Natal
  - Aliwal Shoal Medical and Clinical Trials Center, eMkhomazi, KwaZulu-Natal
  - Tiervlei Trial Center, Bellville, Western Cape
  - Canal Walk Clinical Trial Centre, Cape Town, Western Cape
  - Langeberg Clinical Trials, Cape Town, Western Cape
  - Eden Heart Research Centre, Mossel Bay, Western Cape
- South Korea (9):
  - Yonsei University, Wonju Severance Christian Hospital - Pulmonology, Wŏnju, Gang'weondo [Kang-won-do]
  - Seoul National University Bundang Hospital - Pulmonology, Seongnam-si, Gyeonggido [Kyonggi-do]
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon, Incheon Gwang'yeogsi [Inch'n-Kwangyokshi]
  - Korea University Anam Hospital - Pulmonology, Seoul, Seoul
  - Konkuk University Medical Center, Seoul, Seoul
  - Kyung Hee Universtiy Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Severance Hospital, Yonsei University Health System - Pulmonary, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - The Catholic University of Korea, Seoul St. Mary's Hospital - Pulmonology, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Eunpyeong St. Mary's Hospital, Seoul, Seoul Teugbyeolsi
- Spain (17):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario de Bellvitge - Neumología, L'Hospitalet de Llobregat, Barcelona
  - Hospital Sierrallana - Neumologia, Torrelavega, Cantabria
  - C.A.P. Canet de Mar, Canet de Mar, Catalonia
  - Hospital De Jerez De La Frontera, Jerez de la Frontera, Cádiz
  - Hospital San Pedro de Alcántara, Cáceres, Extremadura
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Fundacion Jimenez Diaz, Madrid, Madrid
  - Hospital Universitario La Paz - Neumologia, Madrid, Madrid
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Vithas Xanit International Hospital - Gastroenterology, Benalmádena, Málaga
  - Hospital Quirónsalud Marbella, Marbella, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Clinica Universidad de Navarra - Neumología, Pamplona, Navarre
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario Virgen del Rocio, Seville, Sevilla
  - Hospital Clinico Universitario De Valencia - Neumologia, Valencia, Valencia
- Taiwan (8):
  - KMU Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung
  - National Taiwan University Hospital - Yunlin Branch - Douliou, Kaohsiung City, Kaohsiung
  - Taichung Veterans General Hospital - Chest Medicine, Taichung, Taichung
  - Kuang Tien General Hospital - XiangShang, Taichung, Taichung
  - Chi Mei Medical Center - YongKang - Pulmonary Medicine, Tainan, Tainan
  - Taipei Medical University - Taipei Medical University Hospital - Internal Medicine, Taipei, Taipei
  - Chang Gung Medical Foundation - LinKou Chang Gung Memorial Hospital - Pulmonary, Taoyuan District, Taoyuan
  - National Taiwan University Hospital - Yunlin Branch - Douliou, Douliu, Yunlin
- Thailand (2):
  - Khon Kaen University, Srinagarind Hospital, Khon Kaen, Changwat Khon Kaen
  - Thammasat University Hospital - Pulmonary and Pulmonary Critic, Khlong Luang, Changwat Pathum Thani
- Turkey (Türkiye) (11):
  - T.C. Saglik Bakanligi - Ankara Etlik sehir Hastanesi, Altındağ, Ankara
  - Hacettepe Universitesi Hastaneleri, Altındağ, Ankara
  - Uludag Universitesi (Uludag University), Beşevler, Bursa
  - T.C. Saglik Bakanligi-S.B.U. Bursa Yuksek Ihtisas Egitim ve Arastirma Hastanesi, Yıldırım, Bursa
  - Istanbul Uni Istanbul Tip Fakultesi, Fatih, Istanbul
  - Marmara University Pendik EAH, Pendik, Istanbul
  - T.C. Saglik Bakanligi - Izmir Sehir Hastanesi, Alsancak, İzmir
  - Medical Park Kocaeli Hastanesi, Köseköy, Kocaeli
  - Inonu Uni. Turgut Ozal Tip Merkezi, Malatya, Malatya
  - Ozel Medical Park Samsun Hastanesi, Samsun, Samsun
  - Karadeniz Teknik Uni Farabi Hastane, Trabzon, Trabzon
- Ukraine (11):
  - KNP "Cherkaska oblasna likarnia", Cherkasy, Cherkasy Oblast
  - KNP"Ts inf.zakhv.Iv-Frank.obl.rady", Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Uzh.miska bahatoprofilna klin.lik., Úzhgorod, Ivano-Frankivsk Oblast
  - MTs "Universalna klinika "Oberih", Kyiv, Kyiv Oblast
  - DU "NNTs im. Yanovskoho", Kyiv, Kyiv Oblast
  - Klin.likarnia na zal.transporti №2, Kyiv, Kyiv Oblast
  - DU "NNTs im. Yanovskoho", Kyiv, Luhansk Oblast
  - MTs "Klinika Hospodarskykh", Ternopil, Ternopil Oblast
  - Medychnyi tsentr "Puls", Vinnytsia, Vinnytsia Oblast
  - Lik.z nevidkl. staniv ta ekstr.dop., Uzhhorod, Zakarpattia Oblast
  - KNP "Likarnia №1" Zhytom.misk.rady, Zhytomyr, Zhytomyr Oblast
- United Kingdom (22):
  - Bioluminux Clinical Research, Milton Keynes, Bedfordshire
  - Synexus Midlands Clinical Research Centre, Edgbaston, Birmingham
  - Velocity Clinical Research - High Wycombe, High Wycombe, Buckinghamshire
  - Royal Primary Care - Ashgate, Chesterfield, Derbyshire
  - Ashburton Surgery, Newton Abbot, Devon
  - Velocity Romford, Romford, Essex
  - NHS Greater Glasgow & Clyde - Gartnavel General Hospital - Respiratory, Glasgow, Glasgow City
  - Panthera Biopartners - Glasgow, Glasgow, Glasgow City
  - Panthera Biopartners - Preston, Preston, Lancashire
  - Leeds Teaching Hospitals NHS Trust - St James' University Hospital, Leeds, Leeds
  - FutureMeds Wirral, Metropolitan Borough of Wirral, Liverpool
  - Panthera Biopartners - North London, Enfield, London
  - Medicines Evaluation Unit, Manchester, Manchester
  - Panthera Biopartners - Manchester, Rochdale, Manchester
  - Lakeside Healthcare, Corby, Northamptonshire
  - Futuremeds - Glasgow, Glasgow, Scotland
  - Panthera Biopartners Sheffield 3 Skye Edge Avenue, Sheffield, Sheffield
  - NHS Tayside - Ninewells Hospital, Dundee, United Kingdom
  - FutureMeds - Newcastle, Newcastle, United Kingdom
  - Royal Berkshire Hospital, Reading, United Kingdom
  - Futuremeds -Teesside, Metropolitan Borough of Wirral, Wirral
  - Panthera Biopartners - York, York, York
- Vietnam (2):
  - University Medical Center of Ho Chi Minh City, Ho Chi Minh City, Ho Chi Minh, Thanh Pho [Sai Gon]
  - Nhan Dan Gia Dinh Hospital, Ho Chi Minh City, Ho Chi Minh, Thanh Pho [Sai Gon]

IPD SHARING:
Plan to Share IPD: No